CLINICAL TRIAL: NCT06701045
Title: Prevalence of Malnutrition and Frailty Among the Urban Community Elderly in Bandung
Status: Completed | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Istingadah Desiana, dr., SpKFR, Ger(K), FIPM(USG), Principal Investigator, Universitas Padjadjaran
Other Study IDs: IKFR-202411.01
Record Dates: First submitted 2024-11-13; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Frail Elderly
Keywords: frail; elderly; malnutrition; community
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elderly living in community: The inclusion criteria were domicile in Bandung City, able to mobilize without assistive devices, able to see and read and willing to participate in the study after informed consent.

SUMMARY:
The goal of this observational study is to learn prevalence of malnutrition and frailty in elderly in Community in Bandung. The main question it aims to answer:

what is the prevalence of malnutrition and frailty in elderly in Bandung community?

DETAILED DESCRIPTION:
The increase in the number and proportion of the elderly population poses various challenges, especially in the health sector. The elderly tend to be more vulnerable to health problems, such as malnutrition and frailty. Data on the prevalence of malnutrition and frailty in the elderly can be used as a basis for taking preventive and treatment measures for both conditions. This study aims to determine the prevalence of malnutrition and frailty in the elderly in the Bandung City community.

Descriptive research with a cross-sectional approach was conducted on 71 elderly participants in the Bandung City community. The sampling method used was consecutive sampling. The study used the Mini Nutritional Assessment-Short Form (MNA-SF) questionnaire to assess malnutrition and the Kihon Checklist (KCL) to assess frailty.

ELIGIBILITY:
Inclusion Criteria:

* age above 60 years old
* domicile in Bandung City
* able to mobilize without assistive devices
* able to see and read
* willing to participate in the study

Exclusion Criteria:

* history of hospitalization within the previous month
* Mini Mental Status Examination ( MMSE ) score < 24

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject were taken form in each district there were a community health center that has an program integrated program specialized for elderly in each subdistrict. We took the subject samples from elderly that regularly visit this subdistrict program.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Frailty | On enrollment
  Frailty is a condition of reduced ability to cope with stressors due to increased vulnerability caused by age-related physiological decline. Frailty score in this study will be measured using Kihon Checklist (KCL) questionnaire that has 24 questions divided into seven categories that are physical strength, nutrition, eating problems, socialization, memory, mood, and lifestyle. The result will bed categorized into not frail (0-3 points), pre-frailty (4-7 points) and frailty (> 8 points).

CONTACTS AND LOCATIONS:
Locations (1):
- Community Health Center, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Small sample size